CLINICAL TRIAL: NCT03879096
Title: Clinical and Functional Variables in the Assessment of Oncology Patient
Brief Title: Clinical and Functional Variables in Oncology
Acronym: Oncolab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Principal Researcher of CTS631 University of Malaga, University of Malaga
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ClubCam
Record Dates: First submitted 2019-03-11; First posted 2019-03-18 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2020-05

CONDITIONS: Cancer, Metastatic; Cancer; Survivorship
Keywords: cancer; oncology; Metastasis; survivors; Exercise Therapy; Therapeutics; Complementary Therapies; fatigue; assesment
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Fatigue | interventions — Exercise Therapy; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): The sample will receive of a Therapeutic Exercise and Education programme
  Interventions: Other: Therapeutic Exercise and Education

INTERVENTIONS:
Other: Therapeutic Exercise and Education — Intervention will consisted of 30 minutes of strength exercises followed by 20 minutes of endurance with aerobic training, individualised based on the evaluations of muscular strength and endurance as well as the determination of the aerobic-anaerobic zone transition. Sessions lasted 1 hour, carried out twice a week, during 12 weeks. This intervention will be complemented by nutritional education.

SUMMARY:
The aim is to analyse the effect of a Therapeutic Exercise and Education programme in several clinical and functional outcomes in cancer patient and survivors

DETAILED DESCRIPTION:
In the oncology field, both patients and survivors have to face several symptoms, like cancer-related fatigue or pain. Cancer patients also have affected quality of life, lower levels of function and they are at higher risk of weight gain following diagnosis. Given the risk of obesity, both exercise and diet play a key role in recovery from cancer.

Hence, the aim of this study is to show the effect of a Therapeutic Exercise and Education programme (TEEP) in clinical and functional, including practical nutritional education in other clinical and functional secondary outcomes in cancer patients and survivors.

Variables included are: body composition, mediterranean-diet adherence, quality of life (QoL) and functional outcomes (limb functionality, physical activity, physical function and handgrip strength). Furthermore, laboratory variables like muscle thickness (ecography) and muscle activity (electromyography) were included.

ELIGIBILITY:
Inclusion Criteria:

* In the case of survivors: Patient who had been surgically treated for their primary tumour with no evidence of recurrence at the time of recruitment. The inclusion of patients undergoing hormonal treatment radiotherapy or antiHER therapy will be allowed.
* In the case of cancer patients: patient who had been dignosed by cancer.

In both cases, all participants have to maintain the minimum physical function to perform exercise in group.

Exclusion Criteria:

* Patients were excluded if they had suffered any cardiovascular event defined as stable or unstable angor, acute pulmonary edema, cardiac rhythm disorders, or syncope of cause not affiliated in the year prior to inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change from Cancer-Related Fatigue (CRF) | Prior and after intervention, an average of 3 months
  The Spanish version of the Piper Fatigue Scale-Revised (PFS-R) will be used
Change from Functional capacity | prior and after intervention, an average of 3 months
  It will be tested by 30-second Sit-To-Stand Test (30-STS), number of repetitions completed.
Change from Upper limb functionality (%) | prior and after intervention, an average of 3 months
  the Spanish version of Upper Limb Functional Index (ULFI) questionnaire will be filled
Change from Lower limb functionality(%) | prior and after intervention, an average of 3 months
  the Spanish version of the Lower Limb Functional Index (LLFI) questionnaire will be filled

SECONDARY OUTCOMES:
Body Composition | prior and after intervention, an average of 3 months
  BMI, basal metabolism, fat/lean mass and water balance will be measured by Tanita TBF-300A
Change from Body Mass Index | prior and after intervention, an average of 3 months
  Body Mass Index calculated based on weight and height as: kilogrames (Kg)/ squared meters (Kg/m2)
Change from Basal Metabolism | prior and after intervention, an average of 3 months
  the number of calories required to keep your body functioning at restm, expressed in Kcal,measured by Tanita TBF-300A
Change from fat mass | prior and after intervention, an average of 3 months
  The fat mass in the total weight of the body, expressed as Kg, measured by Tanita TBF-300A
Change from lean mass | prior and after intervention, an average of 3 months
  The lean mass in the total weight of the body, expressed as Kg, measured by Tanita TBF-300A
Change from water balance | prior and after intervention, an average of 3 months
  Water weight in the total weight of the body, expressed as Kg, measured by Tanita TBF-300A
Change from Physical activity (METS) | prior and after intervention, an average of 3 months
  The International Physical Activity Questionnaire-Short Form (IPAQ-SF) questionnaire will be employed
Change from Handgrip Strength (Kg) | prior and after intervention, an average of 3 months
  Strength will be recorded by Jamar Hydraulic Hand Dynamometer Model SH5001
Change fromQuality of life (self-reported questionnaire) | prior and after intervention, an average of 3 months
  It will be assessed by The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0
Change from specific Breast Cancer Quality of life (self-reported questionnaire) | prior and after intervention, an average of 3 months
  It will be assessed by The European Organization for Research and Treatment of Cancer Breast Cancer-Specific Quality of Life questionnaire (EORTC QLQ-BR23)
Change from Muscle thickness | prior and after intervention, an average of 3 months
  In biceps and cuadriceps muscles, both during relaxation and contraction.
Change from Grip Strength (dynamometry) | prior and after intervention, an average of 3 months
  maximal handgrip strength measured by a The Jamar® Hand Dynamometer (expressed in Kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Antonio Cuesta Vargas, Málaga, Spain

REFERENCES:
- [Background] Quinten C, Maringwa J, Gotay CC, Martinelli F, Coens C, Reeve BB, Flechtner H, Greimel E, King M, Osoba D, Cleeland C, Ringash J, Schmucker-Von Koch J, Taphoorn MJ, Weis J, Bottomley A. Patient self-reports of symptoms and clinician ratings as predictors of overall cancer survival. J Natl Cancer Inst. 2011 Dec 21;103(24):1851-8. doi: 10.1093/jnci/djr485. Epub 2011 Dec 7. PMID 22157640
- [Background] Cuesta-Vargas AI, Buchan J, Arroyo-Morales M. A multimodal physiotherapy programme plus deep water running for improving cancer-related fatigue and quality of life in breast cancer survivors. Eur J Cancer Care (Engl). 2014 Jan;23(1):15-21. doi: 10.1111/ecc.12114. Epub 2013 Aug 16. PMID 23947581
- [Background] Dethlefsen C, Lillelund C, Midtgaard J, Andersen C, Pedersen BK, Christensen JF, Hojman P. Exercise regulates breast cancer cell viability: systemic training adaptations versus acute exercise responses. Breast Cancer Res Treat. 2016 Oct;159(3):469-79. doi: 10.1007/s10549-016-3970-1. Epub 2016 Sep 6. PMID 27601139
- [Background] Cuesta-Vargas AI, Carabantes F, Caracuel Z, Conejo I, Alba E. Effectiveness of an individualized program of muscular strength and endurance with aerobic training for improving germ cell cancer-related fatigue in men undergoing chemotherapy: EFICATEST study protocol for a randomized controlled trial. Trials. 2016 Jan 5;17:8. doi: 10.1186/s13063-015-1143-x. PMID 26732120
- [Background] Cantarero-Villanueva I, Fernandez-Lao C, Diaz-Rodriguez L, Cuesta-Vargas AI, Fernandez-de-las-Penas C, Piper BF, Arroyo-Morales M. The Piper Fatigue Scale-Revised: translation and psychometric evaluation in Spanish-speaking breast cancer survivors. Qual Life Res. 2014 Feb;23(1):271-6. doi: 10.1007/s11136-013-0434-5. Epub 2013 May 22. PMID 23695719
- [Background] Roldan-Jimenez C, Bennett P, Cuesta-Vargas AI. Muscular Activity and Fatigue in Lower-Limb and Trunk Muscles during Different Sit-To-Stand Tests. PLoS One. 2015 Oct 27;10(10):e0141675. doi: 10.1371/journal.pone.0141675. eCollection 2015. PMID 26506612
- [Background] Gerritsen JK, Vincent AJ. Exercise improves quality of life in patients with cancer: a systematic review and meta-analysis of randomised controlled trials. Br J Sports Med. 2016 Jul;50(13):796-803. doi: 10.1136/bjsports-2015-094787. Epub 2015 Dec 30. PMID 26719503
- [Derived] Escriche-Escuder A, Trinidad-Fernandez M, Pajares B, Iglesias-Campos M, Alba E, Garcia-Almeida JM, Roldan-Jimenez C, Cuesta-Vargas AI. Responsiveness of the new index muscular echotexture in women with metastatic breast cancer: an exercise intervention study. Sci Rep. 2022 Sep 7;12(1):15148. doi: 10.1038/s41598-022-19532-7. PMID 36071122
- [Derived] Roldan-Jimenez C, Pajares B, Ruiz-Medina S, Trinidad-Fernandez M, Gonzalez-Sanchez M, Ribelles N, Garcia-Almeida JM, Rios-Lopez MJ, Alba E, Cuesta-Vargas AI. Design and implementation of a standard care programme of therapeutic exercise and education for breast cancer survivors. Support Care Cancer. 2022 Feb;30(2):1243-1251. doi: 10.1007/s00520-021-06470-9. Epub 2021 Aug 31. PMID 34463835